CLINICAL TRIAL: NCT05057481
Title: Reappraisal of Second-line Therapies of Refractory Autoimmune Hemolytic Anemia in Systemic Lupus Erythematosus
Brief Title: Reappraisal of the Therapies of Refractory Autoimmune Hemolytic Anemia in Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Ibrahem Kamel, lecturer in internal medicine department of faculty of medicine,Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17300600
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Autoimmune Hemolytic Anemia; Systemic Lupus Erythematosus
Keywords: autoimmune hemolytic anemia; systemic lupus erythematosus; mycophenolate mofetil
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Lupus Erythematosus, Systemic | interventions — Mycophenolic Acid; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMF arm (Active Comparator)
  Interventions: Drug: Mycophenolate Mofetil 500mg
- Rituximab arm (Active Comparator)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Mycophenolate Mofetil 500mg — MMF 2gram/day orally for 12 weeks
  Arms: MMF arm
Drug: Rituximab — 375 mg/m2 of rituximab given intravenously weekly for 4 weeks.
  Arms: Rituximab arm

SUMMARY:
There is a deficiency in guidelines about the treatment of autoimmune hemolytic anemia in systemic lupus erythematosus (SLE), especially in refractory cases. Mycophenolate mofetil (MMF) showed promising results in those patients but still, the data available are in form of case reports. So, investigators will investigate the efficiency of MMF against a well-established treatment Rituximab in the treatment of refractory autoimmune hemolytic anemia in SLE patients.

DETAILED DESCRIPTION:
There is a deficiency in guidelines about the treatment of autoimmune hemolytic anemia in systemic lupus erythematosus (SLE), especially in refractory cases. Mycophenolate mofetil (MMF) showed promising results in those patients but still, the data available are in form of case reports. So, the investigators will investigate the efficiency of MMF against a well-established treatment Rituximab in the treatment of refractory autoimmune hemolytic anemia in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of erythematosus (SLE) according to The American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) guidelines.
* secondary autoimmune hemolytic anemia (AIHA) that does not respond properly to corticosteroid or when the patients are intolerant to treatment, or refuse standard treatment.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* any contraindication of the used drugs.
* any known hypersensitivity of the used drugs.
* congenital hemolytic anemia.
* chronic renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) proportion | 12 weeks
  CR defined as hemoglobin > 12 g/dL not attributed to transfusion effect and the normalization of hemolytic markers.
partial response (PR) proportion | 12 weeks
  PR defined as hemoglobin 10-12 g/dL or at least ≥ 2 g/dL increase from baseline not attributed to transfusion effect and the normalization of hemolytic markers.
rate of Adverse events | 12 weeks
  rate of occurrence of adverse events of the both drugs

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness | 12 weeks
  Change from baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) sub-scale questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Assiut university, Asyut, Egypt